CLINICAL TRIAL: NCT05130294
Title: A Randomized Controlled Trial Investigating the Efficacy and Safety of Cardio® in Patient With Chronic Obstructive Pulmonary Disease
Brief Title: Unrefined Salmon Oil as Dietary Supplement in Patient With Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated before recruitment began due to administrative decision.
Sponsor: Hofseth Biocare ASA (Industry)
Collaborators: Møre og Romsdal Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CARDIO-COPD; 259935 (Other: Ethics Committee)
Record Dates: First submitted 2021-10-29; First posted 2021-11-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: anti-inflammatory; salmon oil; marine-derived Omega 3; Pulmonary Disease; Chronic Airway Disease; Chronic Obstructive Pulmonary Disease; Obstructive Pulmonary Disease; Lung Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized controlled, double-blinded, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Best Standard of Care + CARDIO® (Active Comparator): 6 gram/day ( 1000 mg per capsule) of unrefined salmon oil, duration of 20 weeks. CARDIO® capsule contains 1000 mg of full spectrum of omega fatty acids, including 21 different fatty acids, with a minimum of 270 mg polyunsaturated fatty acids (PUFA) and10 mg lipopeptides.
  Interventions: Dietary Supplement: CARDIO®
- Best Standard of Care + Placebo (Placebo Comparator): 6 gram/day (1000 mg per capsule) of natural oil, duration of 20 weeks. The placebo is a medium-chain triglyceride (MCT), with triglyceride from natural fatty acid, mainly caprylic- and capric acid.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CARDIO® — CARDIO® is manufactured according to Good Manufacturing Practices for food facilities complying with the Hazard Analysis and Critical Control Points (HACCP) principles.
  The product is intended for use in manufacturing of human food products and human consumption, including food supplements, and have been Generally Recognized as Safe (self-affirmed GRAS). The fresh unrefined salmon oil is produced by Hofseth Biocare ASA
  Arms: Best Standard of Care + CARDIO®
Dietary Supplement: Placebo — MCT oil
  Arms: Best Standard of Care + Placebo

SUMMARY:
Research has over decades showed that marine food carries nutritional characteristics that promote human health. As seen in epidemiological studies and based on in vitro and in vivo studies, it is hypothesized that unrefined salmon oil as dietary supplement have anti-inflammatory effect. However, there is sufficient preliminary data to indicate bioactive compounds effect for clinical use, and further clinical trials investigating effect are needed. This trial will investigate the potential anti-inflammatory effect and reduction in the risk of cardio artery disease in patients diagnosed with chronic obstructive disease, COPD.

DETAILED DESCRIPTION:
This study is a double-blind, placebo-controlled, randomized trial, investigating unrefined salmon oil, CARDIO®, additional to standard care for patients suffering from COPD. The investigational product is an unrefined salmon oil based soft-gel formulation containing 21 different fatty acids (more than 99.1%), lipopeptides (less than 0.9%), antioxidants and other micro metabolites. Research has shown that marine foods carry nutritional characteristics that promote human health, particularly the high intake of long-chain n-3 polyunsaturated fatty acid (n-3 PUFA), eicosapentaeonic acid (EPA), and docosahexaenoic acid (DHA). Cell culture and mouse studies have shown that n-3 PUFAs, such as EPA and DHA, reduce lung leucocyte infiltration and decrease inflammatory cytokines.

Accumulating evidence points to elevated circulating levels of oxidative low-density lipoprotein (ox-LDL) as a key factor that couples COPD with coronary artery disease (CAD). When normal lipoprotein (LDL) becomes oxidized, the structural alteration confers highly pro-inflammatory properties, inducing inflammation and oxidative stress processes central to both COPD and CAD. Ox-LDL is a potent activator of eosinophils, after which the eosinophils appear to mediate chronic inflammation. Based on the literature and studies on the investigational product, the investigators will investigate if CARDIO® can influence eosinophilic inflammation and ox-LDL. This could have positive consequences for improving COPD control and reducing the risk of exacerbations and cardiovascular events. The generalized anti-inflammatory effects and inflammation-resolution promoting effects of unrefined salmon oil might reduce systemic inflammation and benefit COPD patients with co-existing CAD. In this study, the investigators intend to recruit patients with raised oxidative stress represented by patients with serum ox-LDL level at the 25th percentile and above. Therefore, the investigators intend to recruit 20 participants (part 1) with the same inclusion criteria as in part 2, but only measure/analysis serum ox-LDL. The ox-LDL levels derived from part 1 of the study will provide a cut-off level of ox-LDL for patient inclusion into the study part 2. Patient with an ox-LDL value above the 25th percentile will be asked to participate in part 2 of the study. The investigators believe that this will provide the most accurate inclusion of patients to part 2 of the study - the intervention study.

However, clinical trials in humans diagnosed with COPD, have shown varied results investigating n-3 PUFA supplementation. The objective of this study is to evaluate specifically the impact of CARDIO® compared to placebo, on ox-LDL, forced expiratory airflow, blood eosinophils and markers of inflammation in COPD.

Data will be collected by pulmonary function tests (spirometry), blood sample, nutritional log, quality of life questionnaires (CAT), and blood and stool collected for research biobanking. Study intervention period will be 20 weeks, plus 4 weeks post-intervention follow-up, foremost of safety reasons.

As this study is explorative in nature, a sample size which balance the need of statistical power and resource constraints is chosen. The available resources, predetermine those 100 participants, 50 in each arm, can be recruited. Expecting a drop-out rate of about 20% in total (10 subjects per group), and assuming a standard deviation of Ox-LDL of 6 ng/mL the given sample size enables us to detect a mean difference in ox-LDL levels of 3.85 ng/mL. This corresponds to an effect size of 0.64 and shows that the study is reasonably powered. These calculations are done under the standard assumption of power equal to 80% and a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and under treatment for COPD with regular maintenance therapy.
* Postbronchodilator FEV1-FVC ratio less than 0.70 the last 3 months.
* FEV1<90%.
* Current smoker or ex-smoker at least 10 pack-years.
* COPD Assessment Test score level (CAT) ≥10.
* Patients with overlapping COPD and asthma disease may be included.
* Speaks fluent Norwegian.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulation.

Exclusion Criteria:

* Evidence and/or diagnose of clinically significant uncontrolled non-pulmonary disease.

  * Myocardial infarction or stroke within the last 12 months, angina pectoralis diagnosed < 3 months or unstable angina
  * Stage 4 of Congestive Heart Failure according to The New York Heart Association (NYHA) (severe heart failure with poor outcome and decreased survival rate).
  * Cancer diagnosed within the last 12 months (except basal cell carcinoma of the skin), and/or ongoing active cancer therapy.
  * Severe liver disease
  * Severe autoimmune diseases requiring immunosuppressant treatment.
* Pulmonary fibrosis, interstitial lung disease, pulmonary hypertension, sarcoidosis, or significant bronchiectasis.
* Treatment with oral steroid < 1 month prior to baseline visit.
* Oral/intravenous antibiotics < 1 month prior to baseline visit.
* Immunosuppressant therapy such as Cyclosporine and Azathioprine.
* Consumption regularly of fish/krill oil (liquid, capsule, powder) as an oral supplement < 1 month prior baseline visit.
* Known fish or shellfish allergy.
* Participant in any other clinical study.
* Inflammatory bowel disease (Crohn's disease, UC, microscopic colitis), celiac disease, malabsorption, lactose intolerance.
* Severe cognitive impairment where the participants are not able to comply to protocol.
* Any reason why, in the opinion of the investigator, the patient cannot participate, or is not in the patient's best interest.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Level of oxidative low-density lipoprotein (ox-LDL) | Day 0 (baseline) to week 20.
  Across time, change in mean serum level of oxidative low-density lipoprotein (ox-LDL).

SECONDARY OUTCOMES:
Change of C-reactive protein (CRP) | Day 0 (baseline) to week 20.
  Measure mean serum C-reactive protein (CRP) (mg/L), measured between the two treatment groups. Blood samples taken at day 0 (baseline) and 20 week.
Pulmonary airflow measure | Day 0 (baseline) to week 20.
  Mean forced expiratory volume in 1 second (FEV1 ) measured with spirometry at baseline, week 6,12 and 20.
Self-reported measurement in COPD | Day 0 (baseline) to week 20.
  Mean score of COPD assessment test (CAT), measured at week 6,12 and 20.
Pulmonary exacerbation | Day 0 (baseline) to week 20.
  The rate of moderate and severe exacerbations. Moderate exacerbation is defined as use of rescue medication of bronchodilators in combination of antibiotics and/or oral corticosteroids. Severe exacerbation is defined as one that requires hospitalization.
Change of immunregulatory cytokines | Day 0 (baseline) to week 20.
  Mean serum pro-inflammatory cytokines IL-6 and IL-8, measured between the two treatment groups. Blood samples taken at day 0 (baseline) and 20 week.
Rate of composite event | Day 0 (baseline) to 20 week.
  Number of composite score events defined as if one of the following occurs: A worsening of 2 points in self-reported measurement CAT, FEV1 reduction of 100 ml, or Moderate and severe exacerbations. The number of composite score events will be calculated from day 0 (baseline) to 6 weeks, from 6 to 12 weeks, and for 12 to 20 weeks.
Rate of cardiovascular event | Day 0 (baseline) to week 20.
  Number of Major Adverse Cardiovascular Event (MACE) events is defined as if one of the following occurs: Myocardial infarct, Stroke or Cardiovascular death
Concentration of SCFA in stool | Day 0 (baseline) to week 20.
  Determine fecal microbiota composition (16S rRNA) and fecal/plasma metabolome (short-chain fatty acid, SCFA) , measured between the two treatment groups. Stool samples taken at day 0 (baseline) and 20 week.
Change in concomitant medication | Day 0 (baseline) to week 20.
  Any adjustment in concomitant medication during
Change of white blood cells | Day 0 (baseline) to week 20.
  Changes in blood eosinophils (µL), measured between the two treatment groups. Blood samples taken at day 0 (baseline) and 20 week..
Incidence of Treatment-Emergent Adverse Events | Day 0 (baseline) to week 24.
  Safety profile of CARDIO® for each participant randomized to this investigating treatment group. Safety parameters from blood sample of liver function, hemoglobulin, and kidney function will be investigated. The trial will be monitored according to Good Clinical Practice, this to secure the participants safety and well-being. The time frame will be until week 24, four weeks post ended investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Arne L Hoff, MDAssoc.prof, Principal Investigator — More and Romsdal Hospital Trust
Locations (1):
- Hofseth Biocare ASA, Ålesund, More and Romsdal, Norway

IPD SHARING:
Plan to Share IPD: No